CLINICAL TRIAL: NCT00186524
Title: Do Community Cancer Support Groups Reduce Physiological Stress in Women With Primary Breast Cancer?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: California Breast Cancer Research Program (Other); The Wellness Community (Unknown); The Dana Foundation (Other)
Responsible Party: David Spiegel, MD, Stanford University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 4 BB-2901
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Last update posted 2011-03-15 (Estimated); Status verified 2011-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Behavioral: Breast Cancer Support Group

SUMMARY:
Women with primary breast cancer may benefit from participating in supports groups as they cope with treatment and the psychological challenges of survivorship. Studies have documented that these women benefit from support groups run in a university setting; however, no one has documented that they benefit from community cancer support groups. Many community cancer support groups exist and provide service to a large number of women with breast cancer. It is important to know if these groups are providing comparable service to well researched support groups. We conducted this study as the first randomized study of community compared to university-style support groups. Women had a 50/50 chance of being assigned to either a community or a university style support group based on a coin flip. This study took place in two sites The Wellness Community East Bay (Walnut Creek) and San Francisco. Two community groups were studied.

i) This study evaluated the strengths and weaknesses of two community-based support group interventions for breast cancer patients [The Wellness (TWC) and Cancer Support (CSC) Communities, in the San Francisco area]. We compared them with a type of therapy developed in the university setting (Stanford's Supportive-Expressive group therapy), studied which aspects are most effective, and who benefits the most. We compared these women on change in emotional distress, means of coping with cancer, and social and family support. In addition, change in physiological response to stress was measured using saliva samples.

ii) We were able to achieve recruitment for 6 of 8 groups proposed. We randomized 72 women in blocks of 12 taking consecutive women per site until we accrued 12 for each group. Of those, 61 women actually attended groups, of those 46 women to date completed at least one follow-up and were available for analysis for this report. We screened 108 women, 16 who were screened out on initial phone contact, 20 women began to go through our baseline interviews and assessments and either decided not to enroll or dropped out before we could compose a group for the second S.F. randomization. Our final two follow-up assessments for our final group in the East Bay are being conducted right now (8 month) and will be conducted in October, 2002 (12 month) so they are not available for assay or analysis for this final report.

iii) We examined 5 outcome variables for this report and found that women participating in the community groups changed at about the same level over the 4 months of group therapy as the women in the Stanford groups. This was true for depression symptoms, trauma symptoms, social support, self-efficacy, and post-traumatic-growth. These analyses are preliminary until we complete our final follow-up assessments. It is encouraging for the community groups that women benefited at the same rate as they did in the well-researched Stanford groups. Conclusions for this study are somewhat limited because we could not complete the recruitment of our entire sample. However, there is every reason to suppose that community groups are as effective at serving women with primary breast cancer as Stanford's groups though they are based on very different ideas of therapy. It is important to note that all of these groups were led by therapists, and that we may have found other results if the groups had been led by peers or other types of professionals. This study reduces the human and economic cost of breast cancer in California by validating community groups usually offered free to women with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. be > 18 years old
2. be diagnosed with primary breast cancer (Stages I-III, without metastasis or recurrence) within the past 5 years
3. be able to read, speak, and understand English;
4. be < 18 months post treatment; -

Exclusion Criteria:

participation in more than 8 sessions of a support group.

-

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: David Spiegel, M.D., Principal Investigator — Stanford University; Janine Giese-Davis, Ph.D., Study Director — Stanford University; Mitch Golant, Ph.D., Principal Investigator — The Wellness Community; Carol Kronenwetter, Ph.D., Principal Investigator — Cancer Support Community
Locations (3):
- United States (3):
  - Cancer Support Community, San Francisco, California
  - Stanford University, Stanford, California
  - The Wellness Community, Walnut Creek, California

REFERENCES:
- [Background] Cordova MJ, Giese-Davis J, Golant M, Kronnenwetter C, Chang V, McFarlin S, Spiegel D. Mood disturbance in community cancer support groups. The role of emotional suppression and fighting spirit. J Psychosom Res. 2003 Nov;55(5):461-7. doi: 10.1016/s0022-3999(03)00510-5. PMID 14581101